CLINICAL TRIAL: NCT01827683
Title: The Effect of Hyperbaric Oxygen on Patients Suffering From Chronic Pain Syndrome (Fibromyalgia)
Brief Title: Hyperbaric Oxygen and Fibromyalgia: Randomised Prospective Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Principal Investigator, Judith Ben Zvi, medical center, Assaf-Harofeh Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: HBOT-Fibro
Record Dates: First submitted 2011-04-06; First posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Fibromyalgia
Keywords: hyperbaric oxygen; fibromyalgia; chronic pain syndrome
MeSH Terms: conditions — Fibromyalgia | interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyperbaric oxygen therapy group (Active Comparator): hyperbaric oxygen therapy during the first 2 months
  Interventions: Other: Hyperbaric oxygen
- Crossed group (Other): no active intervention during the first 2 months.After 2 months will be crossed to HBOT
  Interventions: Other: Hyperbaric oxygen

INTERVENTIONS:
Other: Hyperbaric oxygen — 8-week, 5 times a week administration of 100% O2 for 90 minutes at a pressure of 2 ATA.

SUMMARY:
The aim of the study is to evaluate the effect of hyperbaric oxygen therapy (HBOT) on patients suffering from chronic pain syndrome (Fibromyalgia).

DETAILED DESCRIPTION:
The study is a prospective, randomized, cross-over trial. Patients will be randomized into two groups (test and control) to receive the HBOT at the beginning of the trial or 2 months afterwards. The control group will receive its treatment after the elapsed two months.

This study will be a prospective, randomized cross over study. After signing a written informed consent, all patients will be invited to a 2 hour examination, including pain sensitivity examination and a series of questionnaires. In addition, prior to the beginning of the treatment all patients will have chest X-ray, neurological examination, cognitive evaluation and brain metabolism evaluation (SPECT scan). A similar evaluation will be done after the 8 weeks, test versus control time period, and another evaluation will be held after 16 weeks. The HBOT procedure will be performed in the hyperbaric chamber at Assaf Harofeh Medical Center, Israel.

The following HBOT protocol will be applied for the treated group: 8-week, 5 times a week administration of 100% O2 for 90 minutes at a pressure of 2 ATA. After 8 weeks the control group, that did not received HBOT, will receive the same HBOT protocols.

At baseline, after 2 months and after 4 months all patients will undergo complete neurologic and pain evaluation and brain SPECT scan (total of 3 evaluation and scan per patient).

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia diagnosed by physical examination of pain sensitivity, by Dolorimeter and finger pressure.

Exclusion Criteria:

* any past hyperbaric oxygen therapy
* chest x-ray pathology which does not allow the income into the hyperbaric chamber.
* middle ear problems.
* patients, who cannot "pump", equals middle ear pressure, effectively.
* patients who suffer from claustrophobia.
* inability or Refusing to sign the Informed Consent Form

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | up to 4 months

SECONDARY OUTCOMES:
Quality of Life | 0,2,4 months
Brain SPECT scan | 0,2,4 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hyperbaric unit, Assaf- Harofe Medical Center, Ẕerifin, Zerifin, Israel

REFERENCES:
- [Derived] Efrati S, Golan H, Bechor Y, Faran Y, Daphna-Tekoah S, Sekler G, Fishlev G, Ablin JN, Bergan J, Volkov O, Friedman M, Ben-Jacob E, Buskila D. Hyperbaric oxygen therapy can diminish fibromyalgia syndrome--prospective clinical trial. PLoS One. 2015 May 26;10(5):e0127012. doi: 10.1371/journal.pone.0127012. eCollection 2015. PMID 26010952